CLINICAL TRIAL: NCT03393221
Title: Enhancing Emotion Regulation Among Overweight and Obese Adolescents Attempting to Lose Weight
Brief Title: Improving Emotion Regulation Skills Among Adolescents Attempting to Lose Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DK108164-01A1 (NIH)
Record Dates: First submitted 2017-12-11; First posted 2018-01-08 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBWC+ER (Experimental): Participants randomized to the Standard Behavioral Weight Control and Emotional Regulation (SBWC+ER) condition receive a 14-session intervention that is comprised of 12 consecutive weekly sessions and 2 booster sessions delivered at weeks 14 and 16. They receive the same information as the Standard Behavioral Weight Control group, but weekly sessions also include elements of TRAC, and it is designed to help teach emotion regulation skills to decrease overeating and sedentary behaviors and increase the likelihood of maintaining diet and exercise behaviors that are taught as part of SBWC interventions.
  Interventions: Behavioral: ER; Behavioral: SBWC
- SBWC (Active Comparator): Participants randomized to the Standard Behavioral Weight Control (SBWC) condition receive a 14-session intervention that is comprised of 12 consecutive weekly sessions and 2 booster sessions delivered at weeks 14 and 16. The intervention includes a dietary plan, a fitness plan, behavioral weight control management that includes self-monitoring, goal-setting, stimulus control strategies, and planning, as well as parental involvement.
  Interventions: Behavioral: SBWC

INTERVENTIONS:
Behavioral: ER — Emotion regulation content
  Arms: SBWC+ER
Behavioral: SBWC

SUMMARY:
While the prevalence of overweight and obesity among children and adolescents has plateaued, national data indicate that approximately 35% of children and adolescents continue to struggle with overweight/obesity. While considerable attention has been given to comprehensive behavioral interventions to address obesity in children, there is less empirical evidence demonstrating efficacy of interventions with adolescents. Additionally, there is great variability and limited impact of adolescent weight control interventions which may be attributable to the failure of these interventions to explicitly address emotion regulation abilities that are necessary for weight loss. Notably, adolescents with poorer general emotion regulation have been found to consume more snack/junk food and report greater amounts of sedentary behavior. Poor emotion regulation among adolescents has also been associated with more rapid weight gain and greater BMI. This project adapts a previously validated Emotion Regulation intervention (TRAC) for at-risk adolescents, targeting sexual risk reduction, to focus on weight loss among a sample of overweight and obese adolescents (ages 12 to 18). While sexual risk and weight management are distinct health behaviors, this same model of emotion regulation could be applied to overweight/obese adolescents attempting to lose weight. In fact, data from overweight/obese adolescents attending a past outpatient weight management program (N=124) indicate that 82% of these youth report emotion regulation scores that are comparable to youth with significant mental health problems. Furthermore, higher levels of emotional dysregulation was associated with greater BMI within this same sample. These data suggest that emotion regulation is related to health decision making and will be relevant to the majority of overweight/obese adolescents seeking to lose weight. The current study will be carried out across Phase 1a and 1b. During Phase 1a, the initial acceptability and feasibility of the adapted intervention (HEALTH TRAC) with eight adolescents in an open pilot trial will be evaluated. During Phase 1b, 48 adolescents between the ages of 13-17 years will be randomized to receive either the HEALTH TRAC or standard behavioral weight control intervention (SBWC) and examine the impact on emotion regulation abilities and BMI status over an eight-month period. The information gained in this project will improve understanding of strategies to improve weight loss outcomes among overweight/obsess adolescents and how improving emotion regulation abilities can enhance these interventions.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years of age
* > 85th percentile for BMI but < a BMI of 50
* speak English
* agree to participation and randomization

Exclusion Criteria:

* they are currently in another weight loss program
* have a medical condition that precludes participation in physical activity or adherence to dietary recommendations
* are developmentally delayed such that the intervention will not be appropriate
* are in treatment for a major psychiatric disorder.
* cannot understand English

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
BMI decrease | baseline, 4 months, and 8 month follow up
  A significant decrease in participant BMI due to weight loss

SECONDARY OUTCOMES:
Emotion Regulation | baseline, 4 month, and 8 month follow up
  Difficulties in Emotion Regulation Scale (DERS)- a 36-item questionnaire designed to assess multiple aspects of emotion regulation (scale: 1 strongly disagree- 5 strongly agree). Measure yields a total score as well as six scales derived through factor analysis: (1. Nonacceptance of emotional response, 2. Difficulties engaging in goal directed behavior [goals], 3. Impulse control difficulties [impulse], 4. Lack of emotion awareness [awareness], 5. Limited access to emotion regulation strategies [strategies] 6. Lack of emotional clarity [clarity] ).
Emotion Regulation Strategy Usage | baseline, 4 month, and 8 month follow up
  Emotion Regulation Behavior Scale (ERBS)- assesses use of emotion regulation strategies taught in intervention. items include "in the last week, when you were having a strong feeling (e.g., sad, upset, etc.) how often did you...get away from whatever was causing your feeling?..."participants respond on a scale of 1 (never) to 5 (all the time) across 8 items, with higher scores indicating more regulatory behaviors (range: 8-40)
Emotion Regulation | baseline, 4 month, and 8 month follow up
  Affect Dysregulation Scale (ADS)- 24 item scale adapted from the clinician-rated Affect Regulation and Experience q-sort questionnaire, modified with 6-items used to assess frequency of difficulty with affect regulation on 4-point Likert, with higher scores indicating more difficulty with affect (range: 6-36)
Emotion Regulation | baseline, 4 month, and 8 month follow up
  Toronto Alexithymia Scale (TAS)- "20 item instrument that is one of the most commonly used measures of alexithymia. Alexithymia refers to people who have trouble identifying and describing emotions and who tend to minimize emotional experience and focus attention externally.
  3 subscales: 1-difficulty describing emotions (5 items-2,4,11,12,17), 2- difficulty identifying emotions (7 items-1,3,6,7,9,13,14), and 3- the tendency of individuals to focus their attention externally (8 items-5,8,10,15,16,18,19,20) "
  (Likert scale: 1 completely disagree - 5 completely agree) (Total range: 20-200)
Distress Tolerance | baseline and 4 months
  Behavior Indicator of Resiliency to Distress (BIRD)- Manipulation/measure of distress-tolerance. The first level of the BIRD test lasts 3 minutes. The level begins with a 5 second latency between dot presentations and changes this latency based on performance (correct answers will reduce the latency by 0.5 seconds whereas incorrect answers or non-responses increase the latency by 0.5 seconds). At the conclusion of this level an average latency is calculated to index skill level. The second level lasts five total minutes. Following a brief rest period the final level begins and lasts for 5 minutes. At all points in the final level the participant will have an escape option. The "quit game" on the screen can be clicked at any time. Therefore making the total time for this game roughly 10-15 minutes long. (Amstadter et al, 2011)
Emotion Regulation | baseline, 4 month, and 8 month follow up
  Emotions as a Child scale- "examines parental emotional socialization from both parent and child perspectives across 45-items. This measure generates 5 subscales of emotion socialization including parental encouragement of emotion expression, parental punishing of responses, parental neglect, parental matching, and parental overriding of child's emotions. Reliability of subscales range from .80 to .87"
Emotion Regulation | baseline, 4 month, and 8 month follow up
  Emotion Regulation Checklist (ERC)- "is an instrument for the hetero-evaluation of the level of emotion regulation of children by means of two scales, Emotion Regulation (ER) and Emotional Lability/ Negativity. 24 items that are assessed on a four point Likert scale (1=never, 2=sometimes, 3=often, and 4= almost always). The ERC comprises two scales: one scale contains 8 items to assess ER, while the other scale contains 15 items that measure emotional liability/negativity, including lack of flexibility, emotional activation, reactivity, anger dysregulation, and mood reliability. (L/N α = .96; ER α = .83), and the two scales are signiﬁcantly correlated (r = -.50, p < .001). One single measurement of ER is generated from the overall scores in both sub-scales (α = .89; Shields & Cicchetti, 1997)."
Emotional Eating | baseline, 4 month, and 8 month follow up
  Emotional Eating Scale (EES)- "25 item self report measure used to assess the propensity to cope with negative affect by eating. Subjects rate their desire to eat in response to each emotion on 5 point scale from "1"I have no desire to eat"" through "5"I have a very strong desire to eat""" (Range 25- 125, with higher scores indicating more coping with affect by eating)
Eating Disorders | baseline, 4 month, and 8 month follow up
  Eating Disorder Examination Questionnaire (EDEQ)- " 28 item questionnaire that has 2 additional questions for males and 5 additional questions for females. Used to measure eating disorder psychopathology, with higher scores indicating higher eating disorder psychopathy. Provides a measure of the range and severity of eating disorder features. Also has the ability to generate operational eating disorder diagnoses. Used to screen potential participants [Subscales: Restraint (items 1,2,3,4,5), Eating concern (items 7,9,19,20,21), Shape concern (items 6,8,10,11,23,26,27,28), Weight Concern (8,12,22,24,25) ]
Eating Habits Confidence | baseline to 8 months
  Eating Habits Confidence Questionnaire (EHCQ)- "27-item scale questionnaire asks participants to rate confidence in their ability to adhere to specific dietary behaviors. Response set consisted of a 5 point-linkert type scale ranging from 1, ""I know I cannot"" to 5, ""I know I can."" Possible scores of this survey range from 27 to 135, with higher scores indicating higher self-efficacy.
Eating Behavior | baseline, 4 months, and 8 months
  Eating Behaviors Inventory- "Instrument for assessing behaviors that have been theoretically implicated in weight loss (self monitoring of food intake and of weight, refusing offers of food, eating at only one place, shopping from a list) 30 items are included that are each rate with a 5 point scale according to how often it was true for the respondent. Items were scored such that the higher scores always reflected more appropriate eating patterns." (Total range: 30- 150)
Accelerometer (physical activity) | baseline and 4 months
  Majority of studies say at least 5 days per week for at least 8 hours per day to receive accurate data on PA. Device used to measure physical activity using criteria such as time spent in activities performed for various intensities and for the prediction of energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hadley, PhD, Principal Investigator — University of Oregon
Locations (1):
- Coro Building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hadley W, Houck C, Barker D, Wickham B, Bogner J, Jelalian E. Preliminary Impact of an Adapted Emotion Regulation Intervention for Adolescents with Overweight and Obesity Attempting to Lose Weight. J Dev Behav Pediatr. 2020 Dec;41(9):706-715. doi: 10.1097/DBP.0000000000000837. PMID 32740283